CLINICAL TRIAL: NCT07362615
Title: An AI-Assisted Art Therapy Co-Creation Intervention for Symptom Burden, Anxiety, and Emotional Regulation in Pediatric Chemotherapy Patients: A Randomized Controlled Trial
Brief Title: An AI-Assisted Art Therapy Co-Creation Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Hazal Ozdemir Koyu, Dr. Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-2254
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer Chemotherapy-Related Symptoms Anxiety
Keywords: pediatric oncology; chemotherapy; AI-assisted intervention; Digital art therapy

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group randomized controlled design. Eligible participants will be randomly assigned in a 1:1 ratio to either the intervention group, which will receive an AI-assisted interactive art-based co-creation program in addition to standard care, or the control group, which will receive standard care alone. Participants will remain in their assigned groups throughout the study, and outcomes will be assessed before and after the four-day intervention period.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants and intervention providers cannot be blinded. However, outcome assessment will be performed by a researcher who is blinded to group allocation. The outcome assessor will not be involved in the intervention delivery and will be unaware of participants' group assignments to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Received standard care
- Intervention Group (Experimental): Participating in an AI-powered art-based program
  Interventions: Other: AI-based art-based program

INTERVENTIONS:
Other: AI-based art-based program — The intervention is an AI-assisted interactive art therapy co-creation program designed to support symptom management, emotional regulation, and anxiety reduction in pediatric patients undergoing chemotherapy. The program is delivered individually during the first 1-4 days of a new chemotherapy cycle and consists of four consecutive daily sessions, each lasting approximately 20-30 minutes.
  The intervention integrates artificial intelligence-generated visual content with child-led artistic expression. In each session, the child interacts with an AI system to generate visual images based on predefined therapeutic themes and personal emotional input. The child then actively completes and personalizes the AI-generated images using their own drawings, colors, and symbols, facilitating emotional expression and engagement.
  The four sessions are structured as follows: (1) establishment of a sense of safety and orientation through initial AI-assisted co-created artwork; (2) symbolic represent
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of an AI-assisted interactive art therapy co-creation intervention on symptom burden, state anxiety, and emotional regulation in pediatric patients receiving chemotherapy. The study will be conducted as a parallel-group randomized controlled trial at the Pediatric Hematology-Oncology units of Gazi University Health Application and Research Center between February 2026 and May 2027. A total of 60 children aged 10-18 years who are undergoing a new chemotherapy cycle will be randomly assigned to either an intervention group receiving a four-day AI-assisted art-based program or a control group receiving standard care. Outcome measures will be assessed before and after the intervention period. The study aims to provide evidence on the feasibility and effectiveness of a short-term, technology-assisted psychosocial intervention to support emotional well-being in children undergoing chemotherapy.

DETAILED DESCRIPTION:
Childhood cancer and its treatment are associated with significant physical and psychological symptom burden, particularly during chemotherapy. Children frequently experience multiple concurrent symptoms such as nausea, pain, fatigue, and sleep disturbances, accompanied by heightened anxiety and emotional distress. These challenges highlight the need for brief, feasible, and developmentally appropriate psychosocial interventions that can be integrated into routine clinical care during active treatment.

This study is designed as a parallel-group randomized controlled trial to examine the effects of an AI-assisted interactive art therapy co-creation intervention on symptom burden, state anxiety, and emotional regulation in pediatric chemotherapy patients. The study will be conducted at the Pediatric Hematology-Oncology units of Gazi University Health Application and Research Center between February 2026 and May 2027.

The study population will consist of children aged 10-18 years who have been receiving cancer treatment for at least six months and are in the first 1-4 days of a new chemotherapy cycle. Eligible participants who meet the inclusion criteria and provide written informed consent (from both the child and parent/legal guardian) will be randomly assigned to either the intervention group or the control group using simple randomization. Randomization will be performed by an independent statistician using an online randomization tool.

The intervention group will receive an AI-assisted interactive art-based program delivered over four consecutive days during chemotherapy, with daily sessions lasting approximately 20-30 minutes. The program is structured into four thematic sessions: (1) creating a sense of safety and introduction through co-created visual artwork with AI, (2) symbolic representation of chemotherapy-related symptoms and coping strategies, (3) exploration of social support and relationships, and (4) future-oriented themes focusing on hope and emotional closure. In each session, children will co-create visual content with AI-generated imagery and complete the artwork with their own drawings.

The control group will receive standard clinical care without any additional psychosocial intervention. Outcome measures will be assessed at baseline (prior to the intervention) and after completion of the four-day program. Data collection tools include a demographic information form, the Symptom Screening in Pediatrics Tool (SSPedi), the State Anxiety Inventory for Children, and the Emotion Regulation Scale for Children.

The primary objective of this study is to evaluate whether the AI-assisted interactive art intervention reduces symptom burden and state anxiety and improves emotional regulation compared to standard care. The findings are expected to contribute to the development of innovative, short-term, and clinically applicable psychosocial interventions and to provide evidence regarding the use of AI-assisted art-based approaches in pediatric oncology care.

ELIGIBILITY:
Inclusion Criteria:

* Be between 10 and 18 years of age
* Have been receiving chemotherapy treatment for at least 6 months
* Be between days 1 and 4 of a new chemotherapy cycle
* Be able to communicate in Turkish
* Be clinically stable
* The participant and their parent/guardian must consent to participate in the study and provide written consent

Exclusion Criteria:

* • Severe neurocognitive impairment, severe physical instability, or being under sedation

  * Experiencing a severe traumatic life event unrelated to the disease within the last 6 months
  * Being in the terminal phase clinically
  * Being under clinical observation due to a psychiatric diagnosis
  * Having fatigue, pain, or medical complications that would prevent participation in the intervention

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Emotional Regulation | Baseline (prior to the intervention) and immediately after completion of the 4-day intervention period
  Emotional regulation will be assessed using the Emotion Regulation Questionnaire for Children and Adolescents. This self-report scale evaluates the use of emotional regulation strategies across two subscales: cognitive reappraisal and expressive suppression. The scale consists of 10 items rated on a 5-point Likert scale. Higher subscale scores indicate more frequent use of the corresponding emotional regulation strategy.
Symptom Burden | Baseline (prior to the intervention) and immediately after completion of the 4-day intervention period
  Symptom burden will be assessed using the Symptom Screening in Pediatrics Tool (SSPedi), a validated self-report instrument for children aged 8-18 years undergoing cancer treatment. The scale includes 15 common physical and psychological symptoms experienced during chemotherapy. Each item is rated on a 5-point Likert scale, with total scores ranging from 0 to 60. Higher scores indicate greater symptom burden and distress.
State Anxiety | Baseline (prior to the intervention) and immediately after completion of the 4-day intervention period
  State anxiety will be measured using the State Anxiety Inventory for Children, a 20-item self-report scale designed to assess situational anxiety levels in children and adolescents aged 8-18 years. Items are rated on a 4-point Likert scale, with total scores ranging from 20 to 80. Higher scores reflect higher levels of state anxiety.

SECONDARY OUTCOMES:
Intervention Acceptability | Immediately after completion of the intervention
  Intervention acceptability and participant satisfaction will be assessed using a researcher-developed process evaluation form. Children will rate their perceived comfort, enjoyment, and satisfaction with the intervention on a numeric scale ranging from 0 to 5, with higher scores indicating greater acceptability.

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding the sharing of individual participant data has not yet been made. Any future data sharing will be considered following completion of the study, in accordance with ethical approval, participant consent, and applicable data protection regulations.

REFERENCES:
- [Result] 1. Chen, Y., Chen, X., Li, L., Li, Y., Yan, Q., & Hu, X. (2025). The efficacy of virtual reality-based interventions on pain, anxiety, depression, and quality of life among patients with cancer: a meta-analysis of randomized controlled trials. Cancer Nursing, 10.1097. 2. Çelik, R., Törüner, E. K., Altay, N., & Bayram, D. (2024). The Validity-Reliability Study of Turkish Version of Electronical Symptom Screening Tool (8-18) in SSPedi-Pediatric Patients with Cancer. Clinical and Experimental Health Sciences, 14(3), 827-834. 3. Dupuis, L. L., Vettese, E., Aftandilian, C., Agarwal, V., Baggott, C., Bradfield, S. M., Crellin-Parsons, N., Freyer, D. R., Kelly, K. M., & King, A. A. (2025). Factors Associated With Self-Report Symptom Screening Adherence in Pediatric Cancer Patients. Cancer Medicine, 14(14), e71053. 4. Gerçeker, G. Ö., Bektaş, M., Önal, A., Kudubeş, A. A., & Çeçen, R. E. (2024). The effect of virtual reality distraction and fatigue training on anxiety and fatigue levels in children with cancer: a randomized controlled study. SEMINARS IN ONCOLOGY NURSING, 5. Hinds, P. S., Grossoehme, D. H., & Reeve, B. B. (2023). One Voice Is Good, But More Is Better: Symptom and Toxicity Reporting in Pediatric Oncology. Cancer Nursing, 46(1), 1-2. 6. Hüzmeli, H., Semerci, R., & Kebudi, R. (2024). The effect of therapeutic play on fear, anxiety, and satisfaction levels of pediatric oncology patients receiving chemotherapy. Journal of pediatric nursing, 77, e195-e201. 7. Jibb, L. A., Yu, A., Nanos, S., Malfitano, C., Foran, L., Hunt, K., Malakian, A., Zimmermann, C., Schultebraucks, K., & Pham, N. A. (2025). The Emotion and Symptom-Focused Engagement (EASE) Psychotherapeutic Intervention for Parents of Children With Acute Leukemia: A Feasibility Trial. Psycho-Oncology, 34(11), e70310. 8. Kisecik Sengul, Z., & Kilicarslan, E. (2025). Investigation into the impact of technology-based motivation program applied to children following cancer diagnosis and their families: a r